CLINICAL TRIAL: NCT03514030
Title: Clinic Registry Study of Optic Neuromyelitis Spectrum Disease in China
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-2
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: NMO Spectrum Disorder;Registry Study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- positive: serum AQP4-antibody is positive
  Interventions: Diagnostic Test: serum AQP4-antibody testing method
- negtive: serum AQP4-antibody is negtive
  Interventions: Diagnostic Test: serum AQP4-antibody testing method

INTERVENTIONS:
Diagnostic Test: serum AQP4-antibody testing method — there are different methods of testing serum AQP4-antibody

SUMMARY:
In 1894, Devic first proposed the concept of neuromyelitis optica(NMO). NMO is an inflammatory demyelinating disease that selectively affects the central nervous system of the optic nerve and spinal cord.In 2004, Lennon and other persons found highly specific AQP4（aquaporin 4）antibodies in NMO patients'sera, and further differentiated between NMO and MS, confirming that NMO is an independent disease.At present, NMO has been widely recognized as an idiopathic and severe demyelinating disease of the central nervous system.In 2015, the international NMO diagnostic team developed the diagnostic criteria based on highly specific AQP4 antibodie.Up to now, in China, there is no data on the number of NMOSD patients, the rate of misdiagnosis, the treatment methods, and the prognosis.This study is committed to build China's NMOSD big data platform to provide the basis for diagnosis, treatment and prognosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. more than 14 years old
2. Compliance with the diagnostic standard by the NMO International Diagnostic team in 2015

Exclusion Criteria:

1. less than 14 years old
2. NOT Compliance with the diagnostic standard by the NMO International Diagnostic team in 2015

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are clinically suspected of being NMOSD
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
misdiagnosis rate | 3 years
  misdiagnosis rate of NMOSD

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes